CLINICAL TRIAL: NCT05304351
Title: A Randomized, Observer-Blind, Phase 2 Study To Assess the Safety and Immunogenicity of CRV-101 Vaccine Head-To-Head With SHINGRIX® for the Prevention of Herpes Zoster in Adults Aged 50 Years and Older
Brief Title: Safety and Immunogenicity of CRV-101 Vaccine for the Prevention of Herpes Zoster in Adults Aged 50 Years and Older
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Curevo Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRV-101-101
Record Dates: First submitted 2021-12-07; First posted 2022-03-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Herpes Zoster; Shingles
Keywords: Herpes Zoster; Shingles; Varicella Zoster Virus; Vaccine
MeSH Terms: conditions — Herpes Zoster; Chickenpox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Arm A (Experimental): Investigational Vaccine
  Interventions: Biological: Amezosvatein Antigen High Dose Arm A
- Arm B (Experimental): Investigational Vaccine
  Interventions: Biological: Amezosvatein Antigen Low Dose Arm B
- Arm C (Active Comparator): Active comparator
  Interventions: Biological: Shingrix
- Arm D (Experimental): Investigational Vaccine
  Interventions: Biological: Amezosvatein Adjuvant Dose Arm D
- Arm E (Active Comparator): Active Comparator
  Interventions: Biological: Shingrix
- Arm F (Experimental): Investigational Vaccine
  Interventions: Biological: Amezosvatein Adjuvant Dose Arm F
- Arm G (Active Comparator): Active Comparator
  Interventions: Biological: Shingrix
- Arm H (Experimental): Investigational Vaccine
  Interventions: Biological: Amezosvatein Adjuvant Dose Arm H
- I (Active Comparator): Active Comparator
  Interventions: Biological: Shingrix
- Arm J (Experimental): Investigational Vaccine
  Interventions: Biological: Amezosvatein Adjuvant Dose Arm J
- Arm K (Active Comparator): Active Comparator
  Interventions: Biological: Shingrix
- Arm L (Experimental): Investigational Vaccine
  Interventions: Biological: Amezosvatein Adjuvant Dose Arm L
- Arm M (Active Comparator): Active Comparator
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: Amezosvatein Antigen High Dose Arm A — Suspension for injection administered intramuscularly (IM) in the deltoid region of the non-dominant arm in Month 0 and Month 2 per study schedule
  Arms: Arm A
Biological: Amezosvatein Antigen Low Dose Arm B — Suspension for injection administered intramuscularly (IM) in the deltoid region of the non-dominant arm in Month 0 and Month 2 per study schedule
  Arms: Arm B
Biological: Shingrix — Suspension for injection administered intramuscularly (IM) in the deltoid region of the non-dominant arm in Month 0 and Month 2 per study schedule
  Arms: Arm C; Arm E; Arm G; Arm K; Arm M; I
Biological: Amezosvatein Adjuvant Dose Arm D — Suspension for injection administered intramuscularly (IM) in the deltoid region of the non-dominant arm in Month 0 and Month 2 per study schedule
  Arms: Arm D
Biological: Amezosvatein Adjuvant Dose Arm F — Suspension for injection administered intramuscularly (IM) in the deltoid region of the non-dominant arm in Month 0 and Month 2 per study schedule
  Arms: Arm F
Biological: Amezosvatein Adjuvant Dose Arm H — Suspension for injection administered intramuscularly (IM) in the deltoid region of the non-dominant arm in Month 0 and Month 2 per study schedule
  Arms: Arm H
Biological: Amezosvatein Adjuvant Dose Arm J — Suspension for injection administered intramuscularly (IM) in the deltoid region of the non-dominant arm in Month 0 and Month 2 per study schedule
  Arms: Arm J
Biological: Amezosvatein Adjuvant Dose Arm L — Suspension for injection administered intramuscularly (IM) in the deltoid region of the non-dominant arm in Month 0 and Month 2 per study schedule
  Arms: Arm L

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of amezosvatein (CRV-101), an investigational vaccine compared to Shingrix® for the prevention of herpes zoster in adults aged 50 years and older

DETAILED DESCRIPTION:
In the first part of the trial, participants will be randomized 1:1:1 to amezosvatein high antigen dose (Arm A), amezosvatein low antigen dose (B), or Shingrix (C). In the second part of the trial, participants will be randomized 5:1 to receive amezosvatein adjuvant dose D or Shingrix (E), adjuvant dose F or Shingrix (G), or adjuvant dose H or Shingrix (I). In the third part of the trial, participants will be randomized 3:1 to receive amezosvatein adjuvant dose J or Shingrix (K) or amezosvatein adjuvant dose L or Shingrix (M). Both study vaccines, amezosvatein and Shingrix, will be administered by intramuscular injection on Month 0 and Month 2. Safety, reactogenicity, and immunogenicity analysis will be performed overall and by age group. Participants will be followed for safety, immunogenicity, and herpes zoster cases from Day 0 to the main study end (Month 14), and through the long-term follow up (LTFU) extension period of up to 5 additional years.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Male and non-pregnant female participant must be ≥50 years of age inclusive, at the time of signing the informed consent.

   * Arms A, B, C, J, K, L, and M will enroll participants ≥50 years of age
   * Arms D, E, F, G, H, and I will enroll participants ≥50 to <70 years of age
2. Participants who are healthy as determined by medical evaluation including comprehensive medical history, comprehensive physical examination, vital signs*, and screening laboratory tests conducted no more than 30 days prior to first study injection administration (Day 0).

   • Vital signs within grade 1 on the severity grading scale, excluding temperature, are allowed. If vital sign parameter meets grade 2 criteria, then subject must be excluded. Vital signs may be repeated 3 times after a period of rest as needed if transient abnormal fluctuation is suspected.
3. (Applicable only for arms A through I) Completed an Emergency Use Authorization (EUA) or Conditional Marketing Authorization or licensed initial COVID-19 vaccine series (as applicable) ≥30 days prior to enrollment (i.e., at least 30 days prior to the Day 0 visit).
4. Screening laboratory values [sodium, potassium, blood urea nitrogen (BUN), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), total bilirubin, alkaline phosphatase, creatinine, random glucose, white blood cell count with differential, hemoglobin, and platelet count] must be within normal ranges or considered not clinically significant by the PI.**
5. Negative HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody at screening. If HIV 1/2 antibody is positive, and confirmation testing is negative the participant may be enrolled.
6. Normal urinalysis or, if abnormal, urinalysis determined to be not clinically significant by the PI at screening.**

   * Screening laboratory values that are abnormal but are considered abnormal due to an acute illness or process may be repeated once. Careful consideration regarding enrolling subjects with screening lab values meeting grade 2 severity that are considered not clinically significant must be made as there is less room for fluctuations to increase to gr ade 3 (severe) lab events.
7. A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

   * Is a woman of nonchildbearing potential (WONCBP). OR
   * Is a woman of childbearing potential (WOCBP) and using an acceptable contraceptive method as defined below during the 30 days prior to Day 0 (i.e., the first study vaccine) and is willing to continue to do so during the study until at least 90 days after the last dose of study vaccine, and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relation to the timing of the first dose of study vaccine.
   * A WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the day of each study vaccine (prior to vaccination). If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.

   WONCBP is as defined as
   * Postmenopausal: A postmenopausal state is defined as least 12 months of spontaneous amenorrhea.
   * Permanently sterile: Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, bilateral oophorectomy, and successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year since of the last menses if menopausal.

   WOCBP is defined as

   • Any woman or adolescent who has begun menstruation. Acceptable contraception methods include, but are not limited to, sexual abstinence, monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the participant receiving study product, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing®, and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill").
8. Capable of understanding and giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol prior to any screening procedures.
9. Willing to abstain from donating whole blood or blood derivatives until after Day 84 visit, and within 60 days prior to each study visit after Day 84.
10. Be able and willing to participate in all study visits and be reachable by telephone or personal contact by the study site personnel.
11. Participants who the investigator believes will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits, have regular contact to allow evaluation during the study).
12. Capable of understanding and completing diary card. Arms A, B, and C use electronic diary and require access to web browser. Arms D through M use paper diary

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. History of herpes zoster (shingles).
2. History or presence of acute or chronic illness (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, hematological, metabolic, gastrointestinal, endocrinologic or renal disorders, or uncontrolled hypertension) which in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
3. History of autoimmune disease or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, HIV infection) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation, or to treat autoimmune disorders) that is likely to affect the immune response to vaccination as determined by the PI.
4. Rash, tattoos, or any other dermatological condition that could adversely affect the vaccine injection site or interfere with its evaluation.
5. Abnormal blood pressure >150 mm Hg systolic or >95 mm Hg diastolic prior to first study injection administration (Day 0).***

   *** If abnormal, BP may be repeated up to 3 times after a rest period of 5 minutes between each measurement.
6. History of significant psychiatric illness (including history of suicidal ideation or attempt) with or without current medication.
7. BMI ≥40kg/m2 at screening (where BMI >34.9 kg/m2, clinically-significant abnormal serum glucose at screening determined by the PI, or clinically-significant diseases or medical conditions, as determined by the PI, is exclusionary.)
8. Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study (e.g., life-threatening disease likely to limit survival to less than 4 years).
9. Acute disease and/or fever at the time of enrollment (Day 0).

   1. Fever is defined as body temperature ≥38 °C (100.4 °F); oral acquisition will be the preferred route for recording temperature throughout this study.
   2. Participants with a minor illness (such as mild diarrhea or mild upper respiratory infection) without fever may be enrolled after resolution of the minor illness, at the discretion of the investigator.
10. Immunized with a vaccine against herpes zoster (Zostavax®, Shingrix®, other licensed or investigational HZ vaccine).
11. Prior varicella vaccination at any time.
12. Received any vaccine within 30 days prior to enrollment (Day 0) or received any non-investigational immunizations while on study except for seasonal influenza, pneumococcal vaccines, other vaccines per the ACIP recommendations, or any licensed or emergency use authorization or conditional marketing authorized COVID-19 booster. Administration of these immunizations must not occur until 30 days after the final study vaccination and completion of the Day 84 immunology blood draw and must not occur within the 30 days prior to each on-study immunology blood draw after Day 84. Receipt of any VZV vaccine is prohibited on the study.
13. Use of any medication that, in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
14. (a) Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs (e.g., oral or injected steroids, such as prednisone; high-dose inhaled steroids; biologics (e.g., tumor necrosis factor [TNF] inhibitor, or other cytokine inhibitors within 14 days of Day 0 through Day 84, and within 14 days of each on study immunogenicity blood draw after Day 84; Exclusionary corticosteroid administration is defined as prednisone >20 mg/day (or equivalent) for any frequency; low-dose inhaled and topical and ocular steroids are allowed; (b) or cytotoxic therapies, such as chemotherapy drugs or radiation, from 180 days prior to enrollment, during the study through Day 421.

    Participants who meet this criterion from 14a and 14b after Day 56, should continue to be followed for safety and immunogenicity but will not be in included in the per protocol population from the date of meeting the criterion.
15. Received a blood transfusion, platelets, plasma, or immunoglobulin 90 days prior to first dose of study vaccine (Day 0) or planned administration of such products during the study.
16. Donated blood products (platelets, whole blood, plasma, etc.) within 60 days prior to enrollment (Day 0).
17. Participation in another experimental protocol which includes the receipt of any investigational products/vaccines or devices within 90 days prior to enrollment (Day 0) in this study, or planned participation in another experimental protocol which includes investigational product/vaccine or device receipt during the study period through D421*. After the D421 visit, participation in another clinical study and with concurrent receipt of another experimental investigational product/vaccine or device is allowed with medical monitor approval. Any other investigational product/vaccine with immune modulating effect which would complicate the assessment of humoral and cellular responses, including investigational vaccines, must not be used 60 days prior to each LTFU extension year visit. Receipt of another experimental VZV vaccine or HSV vaccine is prohibited on the study.

    *Prior to Day 421, concurrent participation in a study which previously included investigational product/vaccine receipt but is no longer receiving investigational products/vaccine, such as in an observational phase of the other study, is allowed.
18. History of previous anaphylaxis or severe allergic reaction to vaccines or sensitivity to any of the study vaccines, or components thereof, or drug or other allergy that, in the opinion of the investigator, contraindicates participation in the study.
19. Known or suspected alcohol or drug abuse within 5 years prior to enrollment (Day 0).
20. ≥20 pack-years for a current smoker or a former smoker at screening.
21. Unlikely to cooperate with the requirements of the study protocol, or deemed unreliable in attending study visits, or otherwise determined by the investigator not to be a good candidate to participate in this study.

[protocol v8.0]

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1516 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2032-03-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited local and systemic signs and symptoms | Day 0-Day 6 for each vaccination timepoint
  Occurrence, severity, and duration of solicited local injection site reactions within 7 days (Day 0-Day 6) following each vaccination. (i.e., pain, redness, swelling)
  Occurrence, severity, and duration of solicited systemic reactions within 7 days (Day 0-Day 6) following each vaccination. (i.e., myalgia, fatigue, headache, chills, fever)
To compare the reactogenicity of amezosvatein to that of the standard 2-dose schedule of Shingrix® | Day 0-Day 6 for each vaccination timepoint
  Comparison of the proportion of participants reporting solicited local and systemic reactogenicity events following each vaccination
Occurrence of unsolicited non-serious adverse events | Day 0-Day 28 following each vaccination
  Occurrence, severity, and relationship to vaccination of unsolicited adverse events within 29 days (Day 0-Day 28) following each vaccination
Occurrence of serious adverse events (SAEs) | Day 0 - Day 421 [Month 14] (as noted in description)
  Occurrence and relationship to vaccination of all serious adverse events (SAE) from after first vaccination (Day 0) to main study end (Day 421 [Month 14])
Occurrence of adverse events (AEs) of special interest | Day 0 - Day 421 [Month 14] (as noted in description)
  Occurrence of any Potential Immune-Mediated Medical Conditions (PIMMCs) from post first vaccination (Day 0) to main study end (Day 421 [Month 14])
  Medically attended adverse events (MAAEs) from post first vaccination (Day 0) to study end (Day 421 [Month 14])
To evaluate safety as measured by hematology and biochemistry parameters | Day 7 and Day 63
  Occurrence, intensity, and relationship to vaccination of clinically significant hematologic and biochemical adverse events at at Day 7 and Day 63
Vaccine protein-specific antibody concentrations (GMC) elicited by vaccination between Month 0 and Month 3 | Month 3
  Assess humoral immune response as determined by Enzyme-linked Immunosorbent Assay (ELISA)
Vaccine Response Rate (≥ 4 fold increase in antibody concentration from pre-vaccination) at Month 3 for arms A, B, and C | Month 3
  • Assess humoral immune response as determined by Enzyme-linked Immunosorbent Assay (ELISA)
To compare the humoral immune response of Shingrix® to amezosvatein | Month 3
  Comparison of humoral response between amezosvatein and Shingrix at Month 3

SECONDARY OUTCOMES:
Fold rise of vaccine protein-specific antibody concentrations elicited in response to vaccination for durability post Month 3 | Month 3
  • Assess humoral immune response as determined by Enzyme-linked Immunosorbent Assay (ELISA)
Anti-Varicella Zoster Virus (VZV) neutralizing antibody titer in response to vaccination between Day 0 and Month 3 for arms A, B, and C | Month 3
  To assess the functional humoral immune response to vaccination (sub-study)
Frequency of vaccine protein-specific CD4+ T cells expressing at least 2 activation markers in response to vaccination between Month 0 and Month 3 for arms A, B, and C | Month 3
  To assess the cell-mediated immunity (CMI) immune response to vaccination as determined by intracellular cytokine staining (ICS)
To compare the frequency of vaccine protein-specific CD4+ T cells expressing at least 2 activation markers of Shingrix® to amezosvatein between Month 0 and Month 3 for arms A, B, and C. | Month 3
  To compare CMI immune response between amezosvatein and Shingrix® at Month 3
CMI Vaccine Response rate (≥ 2-fold increase in the frequency of vaccine protein-specific CD4+ T cell expressing at least 2 activation markers) at Month 3 for arms A, B, and C. | Month 3
  To assess the cell-mediated immunity (CMI) immune response to vaccination as determined by intracellular cytokine staining (ICS)
Vaccine Response Rate (≥ 4 fold increase in antibody concentration from pre-vaccination) at Month 3 for arms D through M | Month 3
  Assess humoral immune response as determined by Enzyme-linked Immunosorbent Assay (ELISA)

OTHER OUTCOMES:
Vaccine protein-specific antibody concentrations elicited by response to vaccination for durability post Month 3 | Month 14, and LTFU up to 5 additional years.
  • Durability of humoral immunogenicity as determined by Enzyme-linked Immunosorbent Assay (ELISA)
Fold rise of vaccine protein-specific antibody concentrations elicited in response to vaccination post Month 3 | Month 14, and LTFU up to 5 additional years.
  • Durability of humoral immunogenicity as determined by Enzyme-linked Immunosorbent Assay (ELISA)
Frequency of vaccine protein-specific CD4+ T cells expressing at least 2 activation markers in response to vaccination for durability post Month 3 | Month 0, Month 14, and in LTFU up to 5 additional years.
  To assess the cell-mediated immunogenicity as determined by intracellular cytokine staining (ICS)
To assess the correlation between vaccine protein-specific Ab concentrations, Anti-VZV neutralizing Ab titer, and frequency of vaccine protein-specific CD4+ T cells expressing >=2 activation markers for each vaccine and correlation across vaccines | Main study (Month 0 - Month 14) and LTFU up to 5 additional years.
  The immunogenicity of amezosvtein alone or compared to Shingrix® will be further evaluated by methods to be determined. Exploratory analyses may include conducting analyses related to furthering the understanding of immunity to VZV and further characterization of the immune responses elicited by amezosvatein and/or in comparison to Shingrix
To evaluate the incidence of clinically confirmed herpes zoster cases | Main study (Month 0 - Month 14) and LTFU up to 5 additional years.
  Occurrence of clinically confirmed herpes zoster cases during the entire main study and LTFU extension period
Frequency of vaccine protein-specific CD4+ T cells expressing at least 2 activation markers in response to vaccination between Month 0 and Month 3 for arms J, K, L, and/or M for dose selected for further development | Month 3
  To assess the cell-mediated immunity (CMI) immune response to vaccination as determined by intracellular cytokine staining (ICS)
To compare Shingrix® to amezosvatein on the frequency of vaccine protein-specific CD4+ T cells expressing at least 2 activation markers between Month 0 and Month 3 for arms J, K, L, and/or M for dose selected for further development | Month 3
  To compare CMI immune response between amezosvatein and Shingrix® at Month 3
CMI Vaccine Response rate (≥ 2-fold increase in the frequency of vaccine protein-specific CD4+ T cell expressing at least 2 activation markers) at Month 3 for arms J, K, L, and/or M for dose selected for further development | Month 3
  To assess the cell-mediated immunity (CMI) immune response to vaccination as determined by intracellular cytokine staining (ICS)
Occurrence of serious adverse events in long term follow up (LTFU) period | LTFU period post Day 421 up to 5 additional years
  Occurrence of serious adverse events in long term follow up (LTFU) period
Occurrence and relationship to vaccination of all serious adverse events (SAE) related or fatal in study participants in LTFU period | LTFU period post Day 421 up to 5 additional years
  Occurrence and relationship to vaccination of all serious adverse events (SAE) related or fatal in study participants in LTFU period
Occurrence of adverse events (AEs) of special interest | LTFU period post Day 421 up to 5 additional years
  Occurrence of any Potential Immune-Mediated Medical Conditions (PIMMCs) in LTFU period

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Shelton, ARNP, Study Director — Curevo Inc; Guy De La Rosa, MD, Study Director — Curevo Inc
Locations (14):
- United States (14):
  - Curevo Investigational Site, Tempe, Arizona
  - Curevo Investigational Site, Coral Gables, Florida
  - Curevo Investigational Site, Tampa, Florida
  - Curevo Investigational Site, Oak Brook, Illinois
  - Curevo Investigational Site, Lenexa, Kansas
  - Curevo Investigational Site, Newton, Kansas
  - Curevo Investigational Site, Lexington, Kentucky
  - Curevo Investigational Site, Las Vegas, Nevada
  - Curevo Investigational Site, Edmond, Oklahoma
  - Curevo Investigational Site, Knoxville, Tennessee
  - Curevo Investigational Site, Austin, Texas
  - Curevo Investigational Site, Dallas, Texas
  - Curevo Investigational Site, Euless, Texas
  - Curevo Investigational Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No